CLINICAL TRIAL: NCT02554630
Title: Novel Mechanisms and Approaches to Treat Neonatal Sepsis: Adjuvant Therapies, Host Microbiome, and Genomic Expression and Functional Capacity of Innate Immune Cells
Brief Title: Novel Mechanisms and Approaches to Treat Neonatal Sepsis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Surgical Infection Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201500447 -N; R01GM097531 (NIH)
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Complication of Prematurity; Immunologic Deficiency Syndromes
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Adjuvants, Pharmaceutic; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Sample Meconium Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preterm Neonate: Neonates of gestational age 24-37 weeks. Blood collection will be performed at the time of a clinically required heelstick or blood draw. Microfluidic techniques, utilizing whole blood, will be employed to characterize the baseline genomic profile and functional capacity of immune cells. Adjuvant drugs will be employed ex-vivo to determine if adjuvant therapies change genomic expression and bolster immune function. Meconium will be collected for microbiome analysis. Clinical outcomes will be recorded from the electronic medical record.
  Interventions: Other: Adjuvant; Other: Blood Collection
- Term Neonates: Neonates of gestational age 37-42 weeks. Blood collection will be performed at the time of a clinically required heelstick or blood draw. Microfluidic techniques, utilizing whole blood, will be employed to characterize the baseline genomic profile and functional capacity of immune cells. Adjuvant drugs will be employed ex-vivo to determine if adjuvant therapies change genomic expression and bolster immune function. Meconium will be collected for microbiome analysis. Clinical outcomes will be recorded from the electronic medical record.
  Interventions: Other: Adjuvant; Other: Blood Collection
- Healthy Adult Control: Healthy Adult aged 18-55 years will undergo a single blood collection by the way of vein puncture. Microfluidic techniques, utilizing whole blood, will be employed to evaluate the genomic profile and functional capacity of immune cells. Adjuvant drugs will be employed ex-vivo to determine if adjuvant therapies change genomic expression and bolster immune function.
  Interventions: Other: Adjuvant; Other: Blood Collection

INTERVENTIONS:
Other: Adjuvant — Blood will be incubated, ex-vivo, with one of the adjuvant therapies or no adjuvant and then, using microfluidic techniques the immune genomic profile and the functional capacity of immune cells will be assessed.
  Other Names: Lippopolysaccaride; Specific toll-like receptor 4 agonist; Non-specific toll-like receptor 4 agonist
Other: Blood Collection — Blood collection will be performed on all groups.

SUMMARY:
Mortality related to neonatal sepsis exceeds 1 million deaths worldwide; the highest risk of mortality is in preterm neonates, especially low birth weight (LBW), and very low birth weight (VLBW) neonates. The estimated cost of caring for these patients is approximately $700 million in the US alone.

In an effort to help mature the neonatal immune system, several adjuvant therapies have been studied; however, none have been implemented in clinical practice. One of the most frequently considered targets for adjuvant therapy is toll-like receptors (TLRs). TLRs detect conserved molecular products of microorganisms (lipopolysaccharide (LPS), and initiate immunity and inflammation. Early adjuvant administration in VLBW infants may be a viable approach to reducing the incidence of early and late sepsis.

This research study will characterize immune genomic expression and functional capacity at the time of birth in both term and preterm neonates and determine what effects, if any, that adjuvants have on this function. Additionally, this study will seek to determine if immune function correlates with certain microbiota.

DETAILED DESCRIPTION:
Blood samples will be collected from three populations: preterm infants, term infants and healthy adult controls. In addition, a collection of meconium (<1mL) from the diaper of these term and preterm neonates;

1. Term neonates (gestational age 37-42 weeks) between birth and 72 hours of life who have blood collected for the following clinical indications:

   a. Blood will be collected at 0-72 hours of life from neonates that are undergoing state metabolic screens or for clinical evaluation jaundice. The sample will be obtained during the standard of care state metabolic screen or for clinical evaluation of jaundice. The neonate will only have an extra drop of blood placed (500-700 micro-liters) in a tube during the heel sticks. Neonates will only have 1 sample drawn throughout the duration of the study.
2. Preterm neonates (gestational age 24-37 weeks) consisting of two populations between birth and 72 hours of life who have blood collected for the following clinical indications:

   1. Blood will be collected at 0-72 hours of life from neonates that are otherwise healthy and do not require additional laboratory testing who are undergoing state metabolic screens or for evaluation of jaundice. The neonate will only have an extra drop of blood placed (500-700 microliters) in a tube during the heel stick. Neonates will only have 1 sample drawn throughout the duration of the study.
   2. A second group of premature neonates will have blood drawn for complications related to prematurity (sepsis work-up). The neonate will only have an extra drop of blood placed (500-700 micro-liters) in a tube during one of these clinical blood draws.
3. Healthy adult controls will have (4milleters) blood collected by way of vein puncture.

For all infants, term and preterm, the following data will be collected at the time of blood collection: gender, gestational age, weight, mechanism of birth (vaginal vs cesarean section), evidence of infectious complication (chorioamnionitis, prolonged rupture of membranes, maternal group B strep colonization, hypoglycemia), use of perinatal antibiotics or steroids, laboratory values available in the electronic medial record (CBC, CMP, Lactic acid, CRP) and Apgar scores will be collected from each patient. Additionally the clinical outcomes of these patients, term and preterm,will be collected until time of discharge but not to exceed 90 days.

ELIGIBILITY:
Preterm and Term neonates 0-72 hours old

Inclusion Criteria:

* Consent to participate in the study

Exclusion Criteria:

* non- survivable condition

Healthy Adult Controls

Inclusion Criteria:

* Consent to participate in the study
* Age >18 years old, <55 years old

Exclusion Criteria:

* Age <18 years old, >55 years old
* Severe pre-existing organ dysfunction
* Oncolytic therapy within 14 days
* HIV positive status
* Current use of chronic steroids

Max Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Preterm neonates 0-72 hours old Term Neonates 0-72 hours old Healthy Adult Controls 18-55 years old
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2016-02; Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Genomic analysis | Day 1
  The genomic profile will be interpreted using Ingenuity Pathway Analysis (IPA) software to make functional predictions. Additionally, a cytokine analysis, and an evaluation for the prevalence of myeloid derived suppressor cells (MDSCs) that have been shown to correlate with poorer outcomes in adult sepsis studies will be performed.
Functional immunologic analysis | Day 1
  Functional capacity will be confirmed directly by observing chemotaxis and quantifying generation of reactive oxygen species (ROS), rate of phagocytosis, and bacterial killing ability. Additionally, a cytokine analysis, and an evaluation for the prevalence of myeloid derived suppressor cells (MDSCs) that have been shown to correlate with poorer outcomes in adult sepsis studies will be performed.

SECONDARY OUTCOMES:
Immune Function Correlation with Clinical Outcomes | 90 days
  The clinical course of these neonates will be followed for incidence of infectious complications including sepsis as evident by culture results. Therefore, allowing the investigators to determine if immunologic deficits present at birth correlate with clinical outcomes.
Ex-vivo Adjuvant Therapies On Immune Function | Day 1
  The implementation of adjuvants in both murine and human models has shown improved function of immune effector cells as well as in clinical outcomes. Adjuvant treatment of mice with TLR agonists stimulates polymorphonuclear leukocytes (PMN) recruitment and function, decreases rates of bacteremia, and increases survival to polymicrobial and gram negative sepsis. Vaccination with Bacillus Calmette-Guerin (BCG) at birth reduces mortality by 40% in LBW infants to sepsis (not tuberculosis) in sub-Saharan Africa. Utilizing an ex-vivo design we will evaluate the changes in immune cell functional capacity.
Ex-vivo Adjuvant Therapies Effect On Immune Cell Genomic Expression | Day 1
  The implementation of adjuvants in both murine and human models has shown improved function of immune effector cells as well as in clinical outcomes. Adjuvant treatment of mice with TLR agonists stimulates polymorphonuclear leukocytes (PMN) recruitment and function, decreases rates of bacteremia, and increases survival to polymicrobial and gram negative sepsis. Vaccination with Bacillus Calmette-Guerin (BCG) at birth reduces mortality by 40% in LBW infants to sepsis (not tuberculosis) in sub-Saharan Africa. Utilizing an ex-vivo design we will evaluate the changes in immune cell genomic expression.
Microbiome Influences Immune Cell Function | Day 1
  Correlated immune deficiencies with differences in the microbiome at the time of birth will be documented by using microbiomic differences present at the time of birth in term vs preterm neonates using Illumina 16s rRNA technology. This system uses highly conserved sequences among bacteria to identify and classify bacterium. The software then provides taxonomic classification to find a microbiomic signature that is specific to immune dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Larson, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Watson RS, Carcillo JA, Linde-Zwirble WT, Clermont G, Lidicker J, Angus DC. The epidemiology of severe sepsis in children in the United States. Am J Respir Crit Care Med. 2003 Mar 1;167(5):695-701. doi: 10.1164/rccm.200207-682OC. Epub 2002 Nov 14. PMID 12433670
- [Background] Lawn JE, Kerber K, Enweronu-Laryea C, Cousens S. 3.6 million neonatal deaths--what is progressing and what is not? Semin Perinatol. 2010 Dec;34(6):371-86. doi: 10.1053/j.semperi.2010.09.011. PMID 21094412
- [Background] Cuenca AG, Wynn JL, Moldawer LL, Levy O. Role of innate immunity in neonatal infection. Am J Perinatol. 2013 Feb;30(2):105-12. doi: 10.1055/s-0032-1333412. Epub 2013 Jan 7. PMID 23297181
- [Background] PrabhuDas M, Adkins B, Gans H, King C, Levy O, Ramilo O, Siegrist CA. Challenges in infant immunity: implications for responses to infection and vaccines. Nat Immunol. 2011 Mar;12(3):189-94. doi: 10.1038/ni0311-189. No abstract available. PMID 21321588
- [Background] Wynn JL, Scumpia PO, Winfield RD, Delano MJ, Kelly-Scumpia K, Barker T, Ungaro R, Levy O, Moldawer LL. Defective innate immunity predisposes murine neonates to poor sepsis outcome but is reversed by TLR agonists. Blood. 2008 Sep 1;112(5):1750-8. doi: 10.1182/blood-2008-01-130500. Epub 2008 Jun 30. PMID 18591384
- [Background] Wynn JL, Levy O. Role of innate host defenses in susceptibility to early-onset neonatal sepsis. Clin Perinatol. 2010 Jun;37(2):307-37. doi: 10.1016/j.clp.2010.04.001. PMID 20569810
- [Background] Yost CC, Cody MJ, Harris ES, Thornton NL, McInturff AM, Martinez ML, Chandler NB, Rodesch CK, Albertine KH, Petti CA, Weyrich AS, Zimmerman GA. Impaired neutrophil extracellular trap (NET) formation: a novel innate immune deficiency of human neonates. Blood. 2009 Jun 18;113(25):6419-27. doi: 10.1182/blood-2008-07-171629. Epub 2009 Feb 12. PMID 19221037
- [Background] Gessler P, Nebe T, Birle A, Haas N, Kachel W. Neutrophil respiratory burst in term and preterm neonates without signs of infection and in those with increased levels of C-reactive protein. Pediatr Res. 1996 May;39(5):843-8. doi: 10.1203/00006450-199605000-00017. PMID 8726239
- [Background] Gentile LF, Nacionales DC, Lopez MC, Vanzant E, Cuenca A, Cuenca AG, Ungaro R, Szpila BE, Larson S, Joseph A, Moore FA, Leeuwenburgh C, Baker HV, Moldawer LL, Efron PA. Protective immunity and defects in the neonatal and elderly immune response to sepsis. J Immunol. 2014 Apr 1;192(7):3156-65. doi: 10.4049/jimmunol.1301726. Epub 2014 Mar 3. PMID 24591376
- [Background] Cuenca AG, Cuenca AL, Gentile LF, Efron PA, Islam S, Moldawer LL, Kays DW, Larson SD. Delayed emergency myelopoiesis following polymicrobial sepsis in neonates. Innate Immun. 2015 May;21(4):386-91. doi: 10.1177/1753425914542445. Epub 2014 Aug 7. PMID 25106654
- [Background] Sweeney SE, Firestein GS. Primer: signal transduction in rheumatic disease--a clinician's guide. Nat Clin Pract Rheumatol. 2007 Nov;3(11):651-60. doi: 10.1038/ncprheum0631. PMID 17968336
- [Background] Kollmann TR, Crabtree J, Rein-Weston A, Blimkie D, Thommai F, Wang XY, Lavoie PM, Furlong J, Fortuno ES 3rd, Hajjar AM, Hawkins NR, Self SG, Wilson CB. Neonatal innate TLR-mediated responses are distinct from those of adults. J Immunol. 2009 Dec 1;183(11):7150-60. doi: 10.4049/jimmunol.0901481. Epub 2009 Nov 16. PMID 19917677